CLINICAL TRIAL: NCT06941779
Title: CuePD: Investigating the Effect of Personalised Auditory Cueing on Gait in Parkinson's Disease
Acronym: CuePD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: North Tyneside General Hospital (Other Government); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CuePD; 327241 (Other: Integrated Research Application System); 24/PR/0684 (Other: Research Ethics Committee)
Record Dates: First submitted 2025-03-31; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease (PD)
Keywords: Wearables; Personalised cueing; Gait retraining

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cueing (Experimental)
  Interventions: Device: Cueing

INTERVENTIONS:
Device: Cueing — Inertial sensors (via a smartphone worn on the lower back) will capture and analyze validated gait-related characteristics (via a gold-standard inertial system worn on both feet). Personalised auditory cues (via smartphone) will be examined for their ability to correct variable gait. To reduce burden on participants (i.e., minimal number of wearable sensors) and to streamline data capture and deliver auditory cues, a single smartphone and a gold standard reference (2 inertial wearables on each foot) will only be used. All devices attached over clothes via belt attachments.

SUMMARY:
Parkinson's Disease (PD) is a major cause of disability, globally. PD affects a person's movement speed, fluency, quality, and ease of walking. PD has the fastest-growing incidence rate, with its prevalence expected to double over the next three decades, currently affecting 10 million people worldwide. PD often leads to disturbances in walking/gait characteristics such as abnormal/variable stride lengths and step times. Those disturbances increase the risk of falls, with about 39% of people with PD (PwPD) experiencing an average of 20.8 falls/year.

Research has examined cueing by leveraging auditory, visual, and tactile cues to normalize variable gait characteristics and improve mobility to reduce falls. Auditory cueing is the most effective at improving gait and most practical to apply in all settings (via headphones) but one size does not fit all when using auditory cueing paradigms i.e., there is a need for personalised approaches to ensure cueing interventions are tailored to the individual and their specific functional limitations. Furthermore, the long-term effectiveness of auditory mechanisms (e.g., metronome-based repetitive beep) suffer from their lack of continuous engagement.

This research project aims to examine personalised auditory cueing to improve gait in PwPD. Inertial sensors will capture and analyze validated gait-related characteristics and personalised auditory cues will be examined for their ability to correct variable gait. To reduce burden on PwPD (i.e., minimal number of wearable sensors) and to streamline data capture and deliver auditory cues, a single smartphone will be used only.

The project involves a multidisciplinary study between Computing and Exercise and Rehabilitation at Northumbria University, testing cueing modalities in a controlled laboratory environment under trained researcher supervision. The study will enrol PwPD, focusing on the ability of personalised auditory cueing to improve gait and PwPD preference of auditory cues.

DETAILED DESCRIPTION:
A researcher will contact identified participants to explain the study further and provide the approved patient information sheet (PIS, via post or email - subject to the potential participant's preference). If after reading the information the potential participant is agreeable, arrangements will be made to book a suitable date and time to visit the Clinical Gait Laboratory, Coach Lane Campus, Northumbria University. Arrangements will be made to ensure the participant has clarity on how s/he can attend the Lab e.g., mode of transport and accessibility.

Upon attending the gait lab informed written consent procedures will be undertaken, then participants (n=60) will be required to answer some demographic questions, such as education level, falls history and activity level. They they will complete pen and paper based clinical assessments such as the Unified Parkinson's Disease Rating scale (UPDRS), Montreal Cognitive Assessment (MoCA), Falls Efficacy Scale-International (FES-I), Falls History Questionnaire, International Physical Activity Questionnaire and Physical Activity questionnaire for Elderly.

Upon completion of the above pen-and-paper tasks, all participants will engage in walking/gait-based tests that assess the effectiveness of a personalised auditory cueing on their gait. All assessments will take place at the Coach Lane Clinical Gait Lab, Northumbria University. During the session, all participants will be asked to wear a smartphone on their person (lower-back via belt attachment), as well as a pair of headphones over their ears and a wearable sensor on each of their feet (the latter are commercial reference standard wearables will be worn on the feet as a gold standard comparison to verify gait data from the smartphone).

Participants will then be asked to perform a series of forward walks around a 25m loop for 1 minute while trying to match their steps to the metronome and musical beats. Walk #1 will determine baseline stepping cadence for each participant. During walks #2-#4 the participant will listen to metronome and musical beats at a +10% increase on the cadence measured during walk #1. After walks #2 and #3, participants will (i) count backwards in their head from 30 to 0 in increments of 1 to disengage psychological responses evoked by each cueing modality and minimize any carryover effects and (ii) perform a 1 min walk with no cue at usual pace.

Specifically, walks and wash-out are:

* Walk 1: Walk for 1-minute at usual pace to determine baseline gait cadence (listening to no sound or no music),

  >> No washout,
* Walk 2: Walk for 1-minute with metronome cueing set at +10% baseline cadence,

  >> Washout (count backwards from 30 to 0 in increments of 1 + 1min walk no cue),
* Walk 3: Walk for 1-minute with instrumental music cueing set at +10% baseline cadence,

  >> Washout (count backwards from 30 to 0 in increments of 1 + 1min walk no cue),
* Walk 4: Walk for 1-minute with vocal music cueing set at +10% baseline cadence.

After the walks, all participants will be asked to answer some questions in the form of a semi-structured interview to explore their experiences of the personalised auditory cueing, administered via a smartphone (System Usability Scale). Goldsmiths Musical Sophistication Index will be used to examine participants' musical experience and skills, and provide valuable insights into the potential of the personalised auditory cueing approach to enhance gait in PwPD. Total time for lab participation is approx 1-hour. The immediate impact of personalised auditory cueing on gait performance in participants will be evaluated based on the collected data and participants' experiences.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk unaided.
* Diagnosis of idiopathic PD, as defined by the UK Brain Bank criteria.
* Score ≥21/30 on Montreal Cognitive Assessment (MoCA) which is used to classify non-demented PD (PD dementia is <21/30).

Exclusion Criteria:

* Non-English speakers
* History of stroke, traumatic brain injury or other neurological disorders (other than PD)
* Acute lower back or lower extremity pain, peripheral neuropathy, and musculoskeletal disorders that would affect tasks.
* Unstable medical condition including cardio-vascular instability in the past 6 months
* Unable to comply with the testing protocol or currently participating in another interfering research project

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gait speed (m/s) | 1 hour
  Average speed of walking in metres per second (m/s) during a 1 minute walk. Measured by the smartphone/IMU via gait-based algorithms located on the lower back.
Step length (m) | 1 hour
  Distance between consecutive steps measured in metres (m). Measured by the smartphone/IMU via gait-based algorithms located on the lower back.
Step time variability | 1 hour
  Coefficient of variation of step time (between consecutive steps). Derrived from the smartphone/IMU via gait-based algorithms located on the lower back. This outcome will determine variability between steps as a proxy for gait stability.
Cadence (steps/minute) | 1 hour
  Calculated as number of steps achieved in one minute (i.e., steps/minute). Derrived from the smartphone/IMU via gait-based algorithms located on the lower back to quantify steps during the 1-min walk.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 15 mins
  Administered as a screening tool to exclude those with cognitive impairment with <21 being a cut-off point for PwPD. The MoCA will be used as a standardised neuropsychological test acknowledged as a valid and efficient tool for the rapid screening of global cognitive dysfunction (Nasreddine, 2005). It is used to examine diverse cognitive domains including attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 40 mins
  Commonly employed to evaluate both motor and non-motor symptoms associated with PD (MDSTF, 2003). This scale consists of four main sections, each targeting a specific area of evaluation. The first part examines non-motor experiences that occur during daily living, while the second part assesses motor experiences during daily living. The third part evaluates motor examination, while the fourth part focuses on assessing complications related to therapy. To determine the severity of the symptoms, the UPDRS is scored based on a total of 195 points, where higher scores suggest increasing levels of disability.
Physical Activity Questionnaire Short Form (IPAQ-SF) | 5 mins
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) will be used to assesses the types of intensity of physical activity and sitting time to estimate total physical activity in MET-min/week and time spent sitting (Craig, 2003).
Physical activity | 5 minutes
  In addition to the IPAQ-SF and to concisely capture physical activity across a range of habitual tasks a secondary physical activity questionnaire will be used. Specifically, the physical activity questionnaire for the elderly with a reference period of 1-year will be used to understand functional household (e.g., cleaning) and community-based activities e.g., shopping (Voorips, 1991).
Falls history | 5 mins
  Falls incidence, cause, location and consequences in the previous 12-months will be assessed by a questionnaire based on recommendations (Lamb 2005, Lord 2007), that leads with the question "In the past year, have you had any fall including a slip or trip in which you lost your balance and landed on the floor or ground or lower level?" (Yardley, 2005).
Falls efficacy | 5 mins
  Used to measure fear of falling in the people with PD (Yardley, 2005). This short, validated measure will assess fear of falling during both basic and demanding activities (physical and social) using a scale from 1 (Not at all concerned) to 4 (Very concerned) across 16 scenarios.
Musical sophistication | 10 mins
  Goldsmiths Musical Sophistication Index (Gold-MSI): A 39-item (scored from 1 to 7) self-report designed to assess musicality across five subscales: active engagement (AE), perceptual abilities (PA), musical training (MT), singing abilities (SA), and emotional response (ER) to music (Müllensiefen, 2014). This tool evaluates and provides the detailed extent and nature of musical experiences and skills, but also provides a broader score on musicality, General Music Sophistication (GMS), ranging from 32 to 126. For this study, the scale will be used to assess if there was a relationship between an individual's general music sophistication and their adherence to the beat of the music cues. Furthermore, the relationship between an individual's subscale results and beat adherence will also be assessed.
System usability | 5 mins.
  System Usability Scale (SUS). This will evaluate perceptions of the app's usability, complexity, and overall satisfaction (Brooke, 2013). The SUS produces a composite score that ranges from 0 to 100, calculated by first adjusting the responses from a set of ten questions. For odd-numbered questions, the process involves subtracting one from each score, whereas for even-numbered questions, the score is subtracted from five, resulting in adjusted values that fall between 0 and 4. These adjusted values are subsequently summed together, and the total is multiplied by 2.5 to derive the final SUS score, with higher scores reflecting superior usability.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Northumbria University, Newcastle
  - North Tyneside General Hospital, North Shields

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brooke J. SUS: a retrospective. Journal of usability studies. 2013;8: 29-40. https://dl.acm.org/doi/10.5555/2817912.2817913
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Voorrips LE, Ravelli AC, Dongelmans PC, Deurenberg P, Van Staveren WA. A physical activity questionnaire for the elderly. Med Sci Sports Exerc. 1991 Aug;23(8):974-9. PMID 1956274
- [Background] Tolosa E, Garrido A, Scholz SW, Poewe W. Challenges in the diagnosis of Parkinson's disease. Lancet Neurol. 2021 May;20(5):385-397. doi: 10.1016/S1474-4422(21)00030-2. PMID 33894193
- [Background] Sweeney D, Quinlan LR, Browne P, Richardson M, Meskell P, OLaighin G. A Technological Review of Wearable Cueing Devices Addressing Freezing of Gait in Parkinson's Disease. Sensors (Basel). 2019 Mar 13;19(6):1277. doi: 10.3390/s19061277. PMID 30871253
- [Background] Rose D, Ott L, Guerin SMR, Annett LE, Lovatt P, Delevoye-Turrell YN. A general procedure to measure the pacing of body movements timed to music and metronome in younger and older adults. Sci Rep. 2021 Feb 5;11(1):3264. doi: 10.1038/s41598-021-82283-4. PMID 33547366
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Mullensiefen D, Gingras B, Musil J, Stewart L. The musicality of non-musicians: an index for assessing musical sophistication in the general population. PLoS One. 2014 Feb 26;9(2):e89642. doi: 10.1371/journal.pone.0089642. eCollection 2014. PMID 24586929
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652
- [Background] Fiorente N, Calabro RS. Music in Parkinson's Disease Rehabilitation: Are We Heading in the Right Direction? Innov Clin Neurosci. 2023 Spring;20(4-6):11-13. PMID 37387705
- [Background] Dotov DG, Cochen de Cock V, Geny C, Ihalainen P, Moens B, Leman M, Bardy B, Dalla Bella S. The role of interaction and predictability in the spontaneous entrainment of movement. J Exp Psychol Gen. 2019 Jun;148(6):1041-1057. doi: 10.1037/xge0000609. PMID 31180717
- [Background] GBD 2016 Parkinson's Disease Collaborators. Global, regional, and national burden of Parkinson's disease, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):939-953. doi: 10.1016/S1474-4422(18)30295-3. Epub 2018 Oct 1. PMID 30287051
- [Background] Allen NE, Schwarzel AK, Canning CG. Recurrent falls in Parkinson's disease: a systematic review. Parkinsons Dis. 2013;2013:906274. doi: 10.1155/2013/906274. Epub 2013 Mar 5. PMID 23533953